CLINICAL TRIAL: NCT02705235
Title: Stress, Coping and Health Behaviors During Pregnancy
Brief Title: Stress, Coping and Health Behaviors in Pregnancy
Status: Completed | Type: Observational
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 0718-15-EP
Record Dates: First submitted 2016-03-05; First posted 2016-03-10 (Estimated); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Pregnancy; Stress; Coping; Health Behaviors
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Stress is an important determinant of pregnancy health behaviors, maternal physiology and maternal-infant health outcomes. The purpose of this study is to explain the relationship between dimensions of lifetime stress and the stress hormone cortisol in pregnant women. Additionally, the study will examine how coping styles help pregnant women to better manage stress and improve their health behaviors to achieve the goal of having a healthy baby.

DETAILED DESCRIPTION:
Health behaviors are important modifiable factors for promoting maternal-infant health during pregnancy, and include behaviors such as diet, exercise, and avoidance of harmful substances. During pregnancy, women are often motivated to improve their lifestyle to achieve positive pregnancy outcomes; however, they may struggle to do so because certain behaviors such as excessive eating, smoking and drinking have become a means for coping with stress. Stress prior to and during pregnancy negatively impacts birth outcomes via complex behavioral and physiologic pathways. From a behavioral perspective, stress diminishes women's engagement in positive health behaviors during pregnancy. From a physiologic perspective, stress affects the regulation of cortisol, a hormone involved in fetal development and timing of delivery. Women use various coping styles to manage stress. It is unknown, however, whether certain coping styles attenuate the negative behavioral and physiologic effects of stress on birth outcomes. Therefore, the purpose of this descriptive, cross-sectional study is to examine the influence of coping styles on stress, physiologic cortisol regulation and health behaviors in a diverse sample of pregnant women (N=55) during 24-28 weeks gestation.

A quantitative design with a qualitative arm will be used to:

1. explain the relationship between cortisol regulation and lifetime stress,
2. determine whether coping styles (active vs. disengaged) moderate the effect of stress on cortisol, health behaviors, and birth outcomes, and
3. describe women's qualitative experience of stress and coping and determine the extent to which the qualitative findings converge with the quantitative findings.

Data will be collected over three prenatal visits during the second half of pregnancy, and will include self-report questionnaires, multiple salivary cortisol sampling, medical record data, a structured stress interview and a semi-structured qualitative interview in a subset of participants (n=12). This study will use an interview-based stress assessment in tandem with physiologic (i.e. cortisol) stress measures in pregnancy. Additionally, the qualitative data will provide a contextual understanding of pregnant women's stress and coping experiences. The research findings will inform the future development and testing of a psychosocial, coping-based intervention to promote positive health behaviors in pregnancy and birth outcomes. Furthermore, this training will provide a solid scientific foundation for the applicant to develop a career as an independent nurse-scientist in maternal-infant health promotion research, under the guidance of an experienced interdisciplinary team of mentors with complementary expertise in stress, coping health behavior, and pregnancy related research. The proposal is consistent with the National Institute of Nursing Research's (NINR) mission to support research that promotes health and prevents disease across the lifespan, builds the scientific foundation for clinical practice, and invests in the training of the next generation of nurse-scientists.

ELIGIBILITY:
Inclusion Criteria:

* Single intrauterine pregnancy at least 20 weeks gestation
* Aged 19 to 45
* Ability to read and speak English
* Able to be reached by telephone or text most days of the week

Exclusion Criteria:

* Receiving or referred for care in the high-risk prenatal clinic
* Have any of the following pregnancy complications or medical issues existing prior to recruitment:

Cervical or uterine abnormalities, renal, hepatic or cardiac disorders, insulin-dependent diabetes, preeclampsia, regular oral steroid use in the month prior to data collection, congenital fetal abnormalities, active placenta previa, blood group isoimmunization, or other disorders/medication use that could affect cortisol levels

* Regular night-shift work or reversed sleep schedule

Ages: 19 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women aged 19 to 45 years old.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2016-01; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Cortisol Awakening Response | 26 weeks gestation
  Participants will collect saliva samples at home by chewing a cotton swab for 1 to 2 minutes. Samples will be collected five times a day for three days. The swab is then placed in a labeled plastic container and stored the container in a home refrigerator. Once returned to the lab, the samples are processed for cortisol awakening response.
Diurnal Slope | 26 weeks gestation
  Participants will collect saliva samples at home by chewing a cotton swab for 1 to 2 minutes. Samples will be collected five times a day for three days. The swab is then placed in a labeled plastic container and stored the container in a home refrigerator. Once returned to the lab, the samples are processed for diurnal slope.
Area Under the Curve (AUC)-Increase | 26 weeks gestation
  Participants will collect saliva samples at home by chewing a cotton swab for 1 to 2 minutes. Samples will be collected five times a day for three days. The swab is then placed in a labeled plastic container and stored the container in a home refrigerator. Once returned to the lab, the samples are processed for index of the sensitivity of the cortisol response to a stressor (AUC-Increase).
Area Under the Curve (AUC)-Ground | 26 weeks gestation
  Participants will collect saliva samples at home by chewing a cotton swab for 1 to 2 minutes. Samples will be collectd five times a day for three days. The swab is then placed in a labeled plastic container and stored the container in a home refrigerator. Once returned to the lab, the samples are processed for total systemic "output" throughout all salivary cortisol measures (AUC-Ground).

CONTACTS AND LOCATIONS:
Overall Officials: Crystal Epstein, PhD, Principal Investigator — University of Nebraska
Locations (1):
- Nebraska Medicine, Omaha, Nebraska, United States